CLINICAL TRIAL: NCT06424665
Title: A PhaseⅠStudy to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of FZ-AD005 in Patients With Advanced Solid Tumors
Brief Title: A Study of FZ-AD005 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F0041-101
Record Dates: First submitted 2024-05-12; First posted 2024-05-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor, SCLC(Small Cell Lung Cancer) or LCNEC (Large Cell Neuroendocrine Carcinoma)
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FZ-AD005 (Experimental)
  Interventions: Drug: FZ-AD005

INTERVENTIONS:
Drug: FZ-AD005 — Every 21 days for 1 cycle. Subjects will receive an intravenous infusion of FZ-AD005 until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.

SUMMARY:
A First-in-Human, Open Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of FZ-AD005 in Patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to give written informed consent;
2. Age ≥ 18 and ≤ 75 years old, male or female;
3. Patients have histological or cytological diagnosis with advanced solid tumors ( especially SCLC or LCNEC);
4. Willingness to provide tumor tissue for testing ;
5. Have measurable lesions defined in RECIST v. 1.1;
6. Expected survival ≥ 3 months;
7. Eastern Cancer Cooperative Group (ECOG) performance status 0-1;
8. Patients of child bearing potential must agree to take contraception during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

1. Patients who have had previous treatment with any anti-DLL3 antibody；
2. Have had other malignant tumors in the past 5 years;
3. Patients who are receiving other anti-tumor treatments within 4 weeks prior to the first dose;
4. Have active CNS (central nervous system) metastasis；
5. Had undergone major surgery or severe trauma within 4 weeks prior to the first dose;
6. Had undergone systemic high-dose steroids within 2 weeks of initiation of study treatment;
7. Patients have psychiatric history;
8. Female patients who are breastfeeding or pregnant;
9. Other reasons that researchers believe are inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The dose limiting toxicity ( DLT) | 21 Days (first cycle)
  To determine the dose limiting toxicities (DLTs) of FZ-AD005
Maximum Tolerable Dose (MTD) | 21 Days (first cycle)
  To determine the maximum tolerated dose (MTD) and/or recommended doses for expansion (RDEs). RDEs will not exceed MTD.
Adverse Events (AEs） | Screening up to study completion, assessed up to 60 months
  To check the numbers of AEs happened during the course of trial.
Objective Response Rate (ORR) | Up to 60 months
  To evaluate the objective response rate (ORR) [Complete Response (CR) + Partial Response (PR)] of FZ-AD005 according to RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival(PFS) | Up to 60 months
  Progression-free survival (PFS) was defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first.
Duration of Response(DOR) | Up to 60 months
  Duration of Response was defined as the duration of overall response measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Overall Survival (OS) | Up to 60 months
  overall survival was defined as the time from the date of the first dose start date to the date of death due to any cause.
Anti Drug Antibody (ADA) | Up to 36 months
  To check the" Anti Drug Antibody" develops in participants against the FZ-AD005 through blood sample
Time to peak (Tmax) | Up to 18 weeks
  To measure the time to reach the maximum contraction of Total Antibody, Free DXd and FZ-AD005 in study participants
Terminal elimination half-life (t1/2) | Up to 18 weeks
  To measure the time of Total Antibody, Free DXd and FZ-AD005 will take to eliminate half of it's concentration from participants.
Maximum observed plasma concentration (Cmax) | Up to 18 weeks
  To measure the maximum concentration participants obtained of Total Antibody, Free DXd and FZ-AD004 in their blood plasma.
Area under the concentration-time curve (AUC 0-∞) from time 0 to infinity | Up to 18 weeks
  To measure the drug profile for absorption, distribution, metabolism and excretion for Total Antibody, Free DXd and FZ-AD005 in participants blood plasma
Time to Cmax (Tmax) | Up to 18 weeks
  To measure the time to reach the maximum contraction of Total Antibody, Free DXd and FZ-AD005 in study participants

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang